CLINICAL TRIAL: NCT07390240
Title: The Effect of Monoallelic Variants in the ALPL Gene on the Natural Course of Hypophosphatasia (HPP) in Children and Adults in Russia
Brief Title: The Effect of Monoallelic Variants in the ALPL Gene on the Natural Course of Hypophosphatasia in Russia
Acronym: ATLANTIS
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8400R00003
Record Dates: First submitted 2025-12-15; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Hypophosphatasia
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
The effect of monoallelic variants in the ALPL gene on the natural course of hypophosphatasia (HPP) in children and adults in Russia (ATLANTIS)

DETAILED DESCRIPTION:
Non-interventional, multi-center, cohort study for evaluation of clinical and patient reported outcomes in routine care settings

ELIGIBILITY:
Inclusion criteria:

1. Age ≥4 to <18 years, or ≥18 years at the time of enrollment;
2. Signed ICF for patients ≥18 years, or legal representatives (parents) of patients aged ≥4 to <18 years;
3. Written informed assent (for patients aged ≥14 to <18 years only);
4. No history of HPP treatment with enzyme-replacement therapy;
5. Diagnosis of HPP confirmed by:

   * reduced alkaline phosphatase (ALP) activity relative to age- and sex-specific reference ranges, confirmed by at least two separate measurements, AND
   * the identification of a monoallelic pathogenic, likely pathogenic, or variant of uncertain significance in the ALPL gene on genetic testing.

Exclusion Criteria:

1. Confirmed conditions presenting with clinical features overlapping with HPP, including but not limited to: cerebral palsy, Duchenne muscular dystrophy, limb-girdle muscular dystrophy (Erb-Roth dystrophy), acquired secondary myopathies of various etiologies;
2. Сurrent participation in any clinical study (patients participating in other non interventional studies may be included);
3. Homozygous or compound heterozygous mutation in the ALPL gene
4. In the opinion of the investigator, the patient is not able to return for follow-up visits or obtain required follow-up studies.
5. Pregnant and breastfeeding women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This multicenter observational study will include 55 paediatric and adult patients newly diagnosed with HPP who carry monoallelic variants in the ALPL gene and are monitored by physicians of various specialties at 5 clinical centers in Moscow and Saint Petersburg, Russian Federation.
  For inclusion to this study, patients should have a documented history of at least 2 reduced alkaline phosphatase (ALP) values relative to age- and sex-specific reference range measured on separate occasions and an HPP diagnosis, but no history of enzyme-replacement therapy. The specific study inclusion and exclusion criteria are described in the sections below.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
(1) Mean age (in full years) at the HPP diagnosis; | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(2) Mean age at the onset of initial HPP symptoms (including separately any, skeletal, and non-skeletal symptoms); | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(3) Proportions of male and female patients | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(4) Proportions of adults and children at baseline (childhood- and adult-onset HPP); | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(5) Proportion of patients with a family history of HPP in a first-degree relative | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(6) Proportions of patients with specific skeletal and non-skeletal manifestation locations/sites affected at baseline: | Day 0 (Visit 1)
  1. Dental;
  2. Skeletal;
  3. Muscular;
  4. Rheumatologic;
  5. Renal;
  6. Respiratory;
  7. Neurologic;
  8. Growth / Development;
  9. Other;
(7) Proportions of patients with history and/or presence of specific skeletal manifestations at baseline: | Day 0 (Visit 1)
  1. Rickets, including all cases, and radiologically confirmed cases;
  2. Skeletal deformities, including all deformities and specific deformities - genu varum, genu valgum;
  3. Osteomalacia;
  4. Osteopenia;
  5. Osteoporosis (for patients aged ≥18 years);
  6. Fractures, including separately:
     all fractures, recurrent metatarsal fractures, all pseudofractures (Looser's zones), atypical femoral fractures, vertebral fractures, wrist fractures, rib fractures, stress fractures of the tibia, and poorly healing fractures (non union); fractures by site: feet, femur (hip), wrist, vertebrae, other bones;
  7. Craniosynostosis;
  8. Bone pain;
  9. Other;
(8) Proportions of patients with history and/or presence of specific dental manifestations at baseline: | Day 0 (Visit 1)
  1. Early nontraumatic loss of primary (deciduous) teeth;
  2. Early atraumatic loss of secondary (adult) teeth;
  3. Periodontal disease;
  4. Other dental abnormalities (separately - abnormal tooth shape and color, enamel thinning/hypoplasia, loss of alveolar bone, enlarged pulp chambers, etc.);
(9) Proportions of patients with history and/or presence of specific muscular manifestations at baseline: | Day 0 (Visit 1)
  1. Muscle weakness;
  2. Enthesopathy;
  3. Low muscle tone;
(10) Proportions of patients with history and/or presence of specific rheumatologic manifestations at baseline: | Day 0 (Visit 1)
  1. Calcium pyrophosphate deposition disease, including separately:
     all cases, pseudogout, and chondrocalcinosis;
  2. Joint pain;
  3. Calcific arthritis and osteoarthritis;
  4. Joint stiffness.
  5. Painful periarticular calcifications of tendons (total and separately - shoulders, elbows, wrists, hips and Achilles' tendons);
(11) Proportions of patients with history and/or presence of specific renal manifestations at baseline: | Day 0 (Visit 1)
  1. Nephrocalcinosis;
  2. Nephrolithiasis (Kidney stones);
  3. Renal impairment / failure (chronic kidney disease);
  4. Other.
(12) Proportions of patients with history and/or presence of specific respiratory manifestations at baseline: | Day 0 (Visit 1)
  1. Frequent respiratory infections;
  2. Chest deformity (e.g., pectus excavatum, kyphosis, scoliosis, flail chest);
  3. Other.
(13) Proportions of patients with history and/or presence of specific neurologic / psychiatric manifestations at baseline: | Day 0 (Visit 1)
  1. Vitamin B6-responsive seizures;
  2. Intracranial hypertension;
  3. Delayed motor milestones;
  4. Cognitive developmental delays;
  5. Waddling gait / difficulty walking;
  6. Depression;
  7. Anxiety;
  8. Attention Deficit/Hyperactivity Disorder;
  9. Insomnia / Poor Sleep Quality;
  10. Other.
(14) Proportions of patients with history and/or presence of other specific manifestations at baseline: | Day 0 (Visit 1)
  1. Fever;
  2. Emesis;
  3. Anorexia;
  4. Polyuria;
  5. Dehydration;
  6. Constipation;
  7. Chronic fatigue;
  8. Other.
(15) Median Standard Deviation Score (SDS) for height at baseline (for patients aged <18 years at the respective timepoints only); | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(16) Proportion of patients with short stature at baseline (SDS for height <-2.0); | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(17) Proportions of patients with other non-specific comorbidities at baseline; | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(18) Proportions of patients with a history and/or presence of specific radiologic signs (X-ray of both hands, posteroanterior view on a single film including the distal forearms) at baseline: | Day 0 (Visit 1)
  1. Metaphyseal rarefaction of bone tissue involving the proximal and middle phalanges;
  2. Epimetaphyseal osteopenia (rarefaction of bone structure) of the forearm bones;
  3. Widened, laminated/striated appearance of the physes of the phalanges and metacarpals, and of the distal epimetaphyseal regions of all visualized bones;
  4. Transverse metaphyseal lines consistent with pathological remodeling in the distal radius and ulna.
(19) Proportions of patients with history and/or presence of specific radiologic signs (radiography of both lower limbs, posteroanterior view on a single full-length film, including the distal lower legs) at baseline: | Day 0 (Visit 1)
  1. Epimetaphyseal osteopenia (rarefaction of bone structure) of the femur, tibia, and fibula;
  2. Transverse striations;
  3. Altered metaphyseal shape: widening;
  4. Epiphyseal hypoplasia;
  5. Flame-shaped metaphyseal changes extending from the epiphyses toward the metaphyses, consistent with hypophosphatasia-related demineralization;
  6. Widening and deformity of the growth plates with a laminated/striated appearance;
  7. Bowing of the long bones of the lower extremities.
(20) Proportions of patients with history and/or presence of specific radiologic signs on standing spine radiographs in anteroposterior and lateral views (preferably full-length) at baseline | Day 0 (Visit 1)
  1. Altered spinal alignment (any, scoliosis, kyphosis);
  2. Altered vertebral shape (any, flattening (platyspondyly), concavity of the upper/lower endplates, wedging);
  3. Altered vertebral structure-osteopenia (of a single vertebra or systemic).
  Children unable to maintain an upright position during radiography may undergo the examination in the supine position in anteroposterior and lateral views).
(21) Proportions of patients with history and/or presence of specific radiologic signs on skull radiographs in anteroposterior and lateral views at baseline: | Day 0 (Visit 1)
  1. Altered contour;
  2. Craniosynostosis;
  3. Altered shape;
  4. Presence of pathological fractures.
(22) Proportions of patients with history and/or presence of specific radiologic signs on foot radiographs in anteroposterior and lateral views (in the presence of clinical signs of a pathological "march" fracture) at baseline: | Day 0 (Visit 1)
  1. Flattening of the transverse arch;
  2. Flattening of the longitudinal arch;
  3. Altered bone structure of the feet, including meta-epiphyseal regions;
  4. Presence of a pathological (march) fracture.
(23) Median Rickets Severity Scale (RSS) at baseline (only for children ≤14 years at the respective timepoints); | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(24) Proportions of patients with history and/or presence of specific laboratory findings at baseline: | Day 0 (Visit 1)
  1. Decreased ALP compared to age- and sex-specific reference values;
  2. Elevated PLP in serum (plasma);
  3. Increased PEA in urine;
  4. Decreased GFR (< 60 ml/min/1.73m2);
  5. Hypocalcemia;
  6. Hypercalciuria;
  7. Decreased PTH;
  8. Increased PTH;
  9. Decreased 25-hydroxyvitamin D;
(25) a Mean and median values of specific laboratory findings at baseline: | Day 0 (Visit 1)
  a) ALP (U/L)
(26) Proportions of patients with specific ALPL gene mutations (for each gene variant); | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(27) Mean and median number of fractures at baseline; | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(28) Mean and median number of dental losses at baseline; | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(29) Mean and median 6-Minute Walk Test (6MWT) distance (m) at baseline (only for patients ≥5 years); | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(30) Proportion of patients with decreased 6MWT distance (m) at baseline (<80% of the predicted norm, only for patients ≥5 years); | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(31) Mean and median Chair-Rise Test time (s) at baseline (only for patients ≥18 years); | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(32) Mean and median Timed Up and Go (TUG) Test time (s) at baseline (only for adults ≥18 years); | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(33) a Mean and median values of specific bioimpedance parameters at baseline | Day 0 (Visit 1)
  a) Total Skeletal Muscle Mass (SMM) (kg);
(34) a Mean and median Rating of Perceived Exertion (RPE) score, based on Borg Scale, during the following specific tests at baseline (when the respective tests have been performed): | Day 0 (Visit 1)
  a) 6MWT;
(35) Mean and median weekly physical activity duration, measured using the International Physical Activity Questionnaire (IPAQ) Diary, at baseline | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(36) Mean and median Pediatric Quality of Life Inventory (PedsQL) score at baseline (only for children <18 years); | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(37) Proportion of patients with different levels of European Quality of Life 5 Dimensions 3-Level (EQ-5D-3L) questionnaire for each of the following dimensions at baseline | Day 0 (Visit 1)
  (1 / 2 / 3): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression (only for adults aged ≥ 18 years);
(38) Mean and median EQ-5D-3L Visual Analogue Scale (VAS) score at baseline (only for adults aged ≥ 18 years); | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(39) Proportion of patients with different Modified Ashworth Scale (MAS) scores (0, 1, 1+, 2, 3, or 4) for each specific muscle / muscle group at baseline: | Day 0 (Visit 1)
  1. Left biceps;
  2. Right biceps;
  3. Paravertebral muscles;
  4. Left femoral quadriceps;
  5. Right femoral quadriceps;
  6. Left calf muscles;
  7. Right calf muscles;
(40) Proportion of patients with clinically significant spasticity (MAS score ≥2 in at least one muscle / muscle group) at baseline; | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(41) Mean and median dynamic component (D) measure based on the modified Tardieu Scale (MTS) on the for each specific muscle / muscle group at baseline (degrees): | Day 0 (Visit 1)
  1. Left biceps;
  2. Right biceps;
  3. Paravertebral muscles;
  4. Left femoral quadriceps;
  5. Right femoral quadriceps;
  6. Left calf muscles;
  7. Right calf muscles;
(42) Proportion of patients with different MTS Resistance scores (0, 1, 2, 3, 4, or 5) for each specific muscle / muscle group at baseline: | Day 0 (Visit 1)
  1. Left biceps;
  2. Right biceps;
  3. Paravertebral muscles;
  4. Left femoral quadriceps;
  5. Right femoral quadriceps;
  6. Left calf muscles;
  7. Right calf muscles;
(43) Proportion of patients with clonus (MTS Resistance score ≥3 in at least one muscle / muscle group) at baseline; | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(44) Proportion of patients with previous hospitalizations due to HPP manifestations at baseline; | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(45) Median number of previous hospitalizations due to HPP manifestations at baseline | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(46) Annualized rate of hospitalizations due to HPP manifestations prior to baseline | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(47) Mean and median duration of previous hospitalizations due to HPP manifestations at baseline | Day 0 (Visit 1)
  In order to achieve the primary objectives, the following variables will be estimated
(48) Proportions of patients with different degrees of disability according to national criteria at baseline | Day 0 (Visit 1)
  1. Group I;
  2. Group II;
  3. Group III;
  4. No disability;
(49) Proportions of patients who had specific previous medical interventions & surgeries at baseline: | Day 0 (Visit 1)
  1. Respiratory support;
  2. Craniotomy;
  3. Other neurosurgical operations;
  4. Dental prostheses;
  5. Fracture fixation/stabilization;
  6. Joint replacement surgeries;
  7. Other orthopedic surgeries;
  8. Orthotics;
  9. Dental implants;
  10. Physical therapy;
(50) Proportions of patients who previously received specific treatments at baseline: | Day 0 (Visit 1)
  1. Pyridoxine;
  2. Antiepileptic medications;
  3. Loop diuretics;
  4. Vitamin D;
  5. Analgesics, including separately:
     Non-steroidal anti-inflammatory drugs (NSAIDs), opioid analgesics, and all analgesics;
  6. Anti-reflux medications;
  7. Teriparatide;
  8. Anti-sclerostin monoclonal antibodies;
  9. Antiresoprtive medications;
  10. Corticosteroids;
  11. Phosphate binders.
(34) b Mean and median Rating of Perceived Exertion (RPE) score, based on Borg Scale, during the following specific tests at baseline (when the respective tests have been performed): | Day 0 (Visit 1)
  b) Chair-Rise Test;
(34) c Mean and median Rating of Perceived Exertion (RPE) score, based on Borg Scale, during the following specific tests at baseline (when the respective tests have been performed): | Day 0 (Visit 1)
  c) TUG Test;
(33) b Mean and median values of specific bioimpedance parameters at baseline | Day 0 (Visit 1)
  b) Lean Body Mass (LBM) (kg);
(33) c Mean and median values of specific bioimpedance parameters at baseline | Day 0 (Visit 1)
  c. Phase angle (degrees)
(25) b Mean and median values of specific laboratory findings at baseline: | Day 0 (Visit 1)
  b) Serum/plasma PLP (ng/ml)
(25) c Mean and median values of specific laboratory findings at baseline: | Day 0 (Visit 1)
  c. Urine PEA (m mol/mol creatinine)
(25) d Mean and median values of specific laboratory findings at baseline: | Day 0 (Visit 1)
  d. GFR (ml/min/1.73m2)
(25) e Mean and median values of specific laboratory findings at baseline: | Day 0 (Visit 1)
  e. Serum calcium (mmol/L)
(25) f Mean and median values of specific laboratory findings at baseline: | Day 0 (Visit 1)
  f. Urine calcium (mmol/24h)
(25) g Mean and median values of specific laboratory findings at baseline: | Day 0 (Visit 1)
  g. Serum PTH (pmol/L)
(25) h Mean and median values of specific laboratory findings at baseline: | Day 0 (Visit 1)
  h. Serum 25-hydroxyvitamin D (ng/ml)

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Research site, Moscow
  - Research site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/